CLINICAL TRIAL: NCT00942929
Title: Lung Function Tests in Adolescents With Anorexia Nervosa
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Bnai Zion Medical Center (Other Government)
Responsible Party: Nogah Kerem, Bnai Zion Medical Centre
Other Study IDs: 48/08
Record Dates: First submitted 2009-07-20; First posted 2009-07-21 (Estimated); Last update posted 2009-07-21 (Estimated); Status verified 2009-07

CONDITIONS: Anorexia Nervosa
Keywords: anorexia nervosa; adolescents; lung function tests; refeeding
MeSH Terms: conditions — Anorexia Nervosa

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Adolescents hospitalized for anorexia nervosa: Adolescent 12-18 years old, fulfilling the DSM IV criteria for anorexia nervosa, hospitalized for medical stabilization and/ or initiation of refeeding
- Controls: Adolescents 12-18 years old without anorexia nervosa hospitalized for reasons other than those involving the respiratory system and with no underlying lung disease

SUMMARY:
The investigators hypothesize that lung function would be adversely affected at the hypocaloric stage of adolescents suffering from anorexia nervosa.

DETAILED DESCRIPTION:
Anorexia Nervosa in adolescents holds adverse effects on different body systems as the cardiovascular, central nervous, endocrine, bone and gastrointestinal systems. There is paucity of information regarding the adverse effects of this tenacious illness on the lungs of adolescents at the hypocaloric stage of their illness. Based on previous clinical observations we postulate that lung function tests would be adversely effected by the hypocaloric nutrition of adolescents with anorexia nervosa and that they may improve during short refeeding in an inpatient setting of a general pediatric ward. To examine our hypothesis we would check lung function by various parameters of adolescents suffering from AN and a control group of adolescents.

ELIGIBILITY:
Inclusion Criteria:

* Adolescents with anorexia nervosa
* Ability to preform lung function tests
* Parents signing informed concent and adolescents signing informed ascent

Exclusion Criteria:

* A history of a lung disease
* Intercurrent lung illness

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Adolescents 12-18 years old hospitalized to a pediatric ward
Sampling Method: Non-Probability Sample
Enrollment: 15 (Estimated)
Dates: Start 2008-09; Study Completion 2009-12 (Estimated)

PRIMARY OUTCOMES:
Lung function tests at admission of adolescents with anorexia nervosa | On addmission to the pediatric ward

SECONDARY OUTCOMES:
Lung function tests at discharge of adolescents with anorexia nervosa | On discharge from the pediatric ward

CONTACTS AND LOCATIONS:
Locations (1):
- Bnai Zion Medical Centre, Department of Pediatrics, Haifa, Israel